CLINICAL TRIAL: NCT04720157
Title: An Open-label, Randomized, Phase III Study Comparing 177Lu-PSMA-617 in Combination With Standard of Care, Versus Standard of Care Alone, in Adult Male Patients With Metastatic Hormone Sensitive Prostate Cancer (mHSPC)
Brief Title: An International Prospective Open-label, Randomized, Phase III Study Comparing 177Lu-PSMA-617 in Combination With Standard of Care (SoC), Versus SoC Alone, in Adult Male Patients With Metastatic Hormone Sensitive Prostate Cancer (mHSPC)
Acronym: PSMAddition
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Alliance Foundation Trials, LLC. (Other); RTOG Foundation, Inc. (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617C12301; 2023-507970-42-00 (Other: EU CTIS)
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Prostatic Neoplasms
Keywords: Lutetium-177 PSMA-617; 177Lu-PSMA-617; Androgen receptor-directed therapy; ARDT; Androgen Deprivation Therapy; ADT; Metastatic Hormone sensitive prostate cancer; mHSPC; Radiographic progression free survival; rPFS; Prostate-specific membrane antigen; PSMA; Gallium-68 PSMA-11; 68Ga-PSMA-11; Radioligand Therapy; RLT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: Patient randomized to SOC arm have an option to crossover to 177Lu-PSMA-617 treatment after rPFS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 177Lu-PSMA-617 (Experimental): Participant will receive 7.4 GBq (+/- 10%) 177Lu-PSMA-617, once every 6 weeks (+/- 1 week) for a planned 6 cycles, in addition to the Standard of Care (SOC); Androgen receptor-directed therapy (ARDT) + Androgen deprivation therapy (ADT) is considered as SOC and treatment will be administered per the physician's order
  Interventions: Drug: 177Lu-PSMA-617; Drug: 68Ga-PSMA-11; Drug: ARDT; Drug: ADT
- Standard of Care (Active Comparator): For participants randomized to Standard of Care arm, ARDT +ADT is considered as SOC and treatment will be administered per the physician's order
  Interventions: Drug: 68Ga-PSMA-11; Drug: ARDT; Drug: ADT

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — administered intravenously once every 6 weeks (1 cycle) for 6 cycles
  Other Names: AAA617
  Arms: 177Lu-PSMA-617
Drug: 68Ga-PSMA-11 — Intravenous dose of approx. 150 Megabecquerel (MBq) at screening and at time of centrally confirmed rPD
Drug: ARDT — Administered orally on a continuous basis as per package insert and guideline
Drug: ADT — ADT are administered as per physician order

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 177Lu-PSMA-617 in combination with Standard of Care (SOC), versus Standard of Care alone, in adult male patients with Metastatic hormone sensitive prostate cancer (mHSPC). In this study, the SoC is defined as a combination of Androgen Receptor Directed Therapy + Androgen Deprivation Therapy. Approximately 1126 patients will be randomized in this study. As of 31-Jan-2024, 1144 participants were enrolled in 20 countries.

DETAILED DESCRIPTION:
In this international, open-label, prospective, phase III study, where approximately 1126 patients with treatment naïve or minimally treated PSMA-positive mHSPC were to be randomized in a 1:1 ratio to receive Standard of Care (SoC) with or without the radioligand 177Lu-PSMA-617.

The primary objective of the study was to determine whether the combination of 177Lu-PSMA-617 + SoC improved radiographic progression free survival (rPFS) over that obtained by administration of SoC alone in mHSPC patients.

The randomization was stratified according to the following three factors: disease volume (high v low), age >= 70 years (yes/no), and on Previous or planned treatment (prostatectomy or radiation) to primary (prostate) tumor (yes/no).

Study duration: approximately 50 months. screening period: after signing ICF, patients were assessed for eligibility and were scanned with 68Ga PSMA-11 to identify PSMA expression status. Following completion of all required screening procedures and verifying participant eligibility, the participant was randomized via the interactive response technology (IRT) system.

Amended protocol v02 included an option for participants to be enrolled into a separate long-term safety follow-up study, and China extension cohort (40 to 60 participants). Amended protocol v03 excluded China extension cohort and added a second 68Ga-PSMA-11 PET/CT scan at rPD.

Prior treatment:

* Up to 45 days of Luteinizing hormone releasing hormone (LHRH) agonist/antagonists was allowed prior to informed consent form (ICF) signature. If patient did not start the ADT prior randomization, ADT started as soon as possible and ideally no later than 2 weeks after randomization.
* Up to 45 days of ARDT was allowed prior ICF signature. If patient did not start the ARDT prior randomization, ARDT started as soon as possible and ideally no later than 2 weeks after randomization. Patients received ARDT as per label instructions.

Randomization period:

The participant was randomized in a 1:1 ratio to receive Standard of Care (SoC) with or without the radioligand 177Lu-PSMA-617.

Treatment period:

Patients randomized to the investigational arm (i.e. SoC+177Lu-PSMA-617): Patients received SoC as per label instructions, after randomization, if not started earlier and in the time frame allowed by the protocol. Patients began 177Lu-PSMA-617 dosing within 14 days after randomization or as soon as possible after the product was received. 177Lu-PSMA-617 is administered at the dose of 7.4 GBq (+/- 10%), once every 6 weeks (+/- 1 week) for a planned 6 cycles.

Patients randomized to the control arm began receiving SoC as per label instructions after randomization, if not started earlier and in the time frame allowed by the protocol.

The primary endpoint of rPFS was assessed by a centralized blinded image review committee (i.e., BIRC) using radiographic images provided by the treating physician.

Participants from both arms also underwent PET/CT scan with 68GaPSMA-11 following Centrally confirmed rPD.

An end of treatment (EOT) visit will be performed when participants permanently discontinue study treatment.

Cross-over period:

After patients randomized to the SoC alone (i.e., control) arm experience radiographic progression (the rPFS event) as confirmed by BIRC, they will be allowed to cross-over to receive 177Lu-PSMA-617 +/- SoC per the discretion of the treating physician. If cross-over to 177Lu-PSMA-617 is selected, then 177Lu-PSMA-617 will be administered with the same dose/schedule as participants who were initially randomized to receive 177Lu-PSMA-617 as described above. Study cross-over participants for whom 177Lu-PSMA-617 is discontinued must have a second End of Treatment (EOT2) visit performed =< 7 days and enter the Post-treatment Follow-up.

Post-Treatment Follow-Up (Safety, Efficacy):

After treatment discontinuation, all participants will be followed for safety with a 30-day safety follow-up visit (FUP) as well as longer term safety follow-up assessments for a period of approximately 12 months.

Participants who discontinue study treatment without having progressive disease confirmed by BIRC, will continue to be assessed for efficacy (efficacy follow-up) during the post-treatment follow-up period until the occurrence of their BIRC-confirmed radiographic disease progression (rPFS) event , or if the total number of protocol-defined rPFS events has occurred triggering the primary analysis, whichever occurs first.

Survival Follow-Up:

After study treatment discontinuation, or post-treatment follow-up period discontinuation, the participant's status will be collected every 90 days (via phone calls) as part of the survival follow-up. Every effort should be made to comply with the survival follow-up schedule and ensure collection of participant survival. The survival follow-up and the study will end when the number of OS events required for final OS analysis will be reached.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Patients must be adults ≥18 years of age
3. Patients must have an ECOG performance status of 0 to 2
4. Patients must have a life expectancy >9 months as determined by the study investigator
5. Patients must have metastatic prostate cancer with histologically or cytologically confirmed adenocarcinoma (current or prior biopsy of the prostate and/or metastatic site)
6. Patients must have evidence of PSMA-positive disease as seen on a 68Ga-PSMA-11 PET/CT scan, and eligible as determined by the sponsor's central reader
7. Patients must have at least one documented metastatic bone and/or soft tissue/visceral lesion documented in the following manners within 28 days prior randomization:

   1. Metastatic disease to the bone (in any distribution) visible on 99Tc-MDP bone scintigraphy on either pre-ADT scans or baseline scans AND/OR
   2. Lymph node metastases of any size or distribution. If lymph nodes are the only site of metastasis, then at least one must be at least 1.5 cm in short axis AND outside of the pelvis AND/OR
   3. Visceral metastases of any size or distribution. If a participant has a history of visceral metastases at any time prior to randomization, he should be coded as having visceral metastases at baseline (i.e., patients with visceral metastases prior to ADT that disappear at baseline will be counted as having visceral metastases and would therefore have high volume disease for stratification purposes).
8. Patients must have adequate organ function:

   * Bone marrow reserve ANC ≥1.5 x 109/L Platelets ≥100 x 109/L Hemoglobin ≥9 g/dL
   * Hepatic Total bilirubin ≤2 x the institutional upper limit of normal (ULN). For patients with known Gilbert's Syndrome ≤3 x ULN is permitted Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3.0 x ULN OR ≤5.0 x ULN for patients with liver metastases
   * Renal eGFR ≥ 50 mL/min/1.73m2 using the Modification of Diet in Renal Disease (MDRD) equation
9. Albumin ≥2.5 g/dL
10. Human immunodeficiency virus (HIV)-infected patients who are healthy and have a low risk of acquired immune deficiency syndrome (AIDS)-related outcomes can participate in this trial
11. Patients must be:

Treatment naïve OR minimally treated with:

* Up to 45 days of luteinizing hormone-releasing hormone (LHRH) agonist /antagonists or bilateral orchiectomy with or without first generation anti-androgen (e.g. bicalutamide, flutamide) for metastatic prostate cancer is allowed prior to ICF signature. If given, first generation anti-androgen must be discontinued prior to start of study therapy or after 45 days whatever happens first.
* If received, prior LHRH agonist/antagonist with or without first generation anti-androgen use in the adjuvant/neo-adjuvant setting must have been discontinued > 12 months prior to ICF signature AND must not have exceeded 24 months of therapy AND must not have shown disease progression within 12 months of completing adjuvant/neo-adjuvant therapy.
* Up to 45 days of CYP17 inhibitor or ARDT exposure for metastatic prostate cancer is allowed prior to ICF signature. No CYP17 inhibitor or ARDT exposure for earlier stages of prostate cancer is allowed.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for inclusion in this study.

1. Participants with rapidly progressing tumor that requires urgent exposure to taxane-based chemotherapy
2. Any prior systemic anti-prostate cancer therapy (with the exception of the drugs listed on inclusion criteria 11), including chemotherapy, Poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitors, immunotherapy or biological therapy (including monoclonal antibodies).
3. Concurrent cytotoxicity chemotherapy, immunotherapy, radioligand therapy, PARP inhibitor, biological therapy or investigational therapy
4. Previous treatment with any of the following within 6 months of randomization: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation. Previous PSMA-targeted radioligand therapy is not allowed
5. Ongoing participation in any other clinical trial
6. Use of other investigational drugs within 30 days prior to day of randomization
7. Known hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical classes
8. Transfusion for the sole purpose of making a participant eligible for study inclusion
9. Participants with CNS metastases that are neurologically unstable, symptomatic, or receiving corticosteroids for the purpose of maintaining neurologic integrity. Participants with epidural disease, canal disease and prior cord involvement are allowed if those areas have been treated, are stable, and not neurologically impaired. Participants with parenchymal CNS metastasis (or a history of CNS metastasis), that have received prior therapy and are neurologically stable, asymptomatic and not receiving steroids for CNS metastases, are allowed, baseline and subsequent radiological imaging must include evaluation of the brain (magnetic resonance imaging (MRI) preferred or CT with contrast).
10. Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, participants with a prior history of malignancy that has been adequately treated and who have been disease free, treatment free for more than 3 years prior to randomization, or participants with adequately treated non-melanoma skin cancer, superficial bladder cancer are eligible.
11. Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, uncontrolled infection, known active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation. Participants with an active documented COVID-19 infection (any grade of disease severity) at time of informed consent may be included only when completely recovered (in accordance with local guidance).
12. Active clinically significant cardiac disease defined as any of the following:

    * NYHA class 3/4 congestive heart failure within 6 months prior to ICF signature unless treated with improvement and echocardiogram or MUGA demonstrates EF > 45% with improvement in symptoms to class < 3.
    * History or current diagnosis of ECG abnormalities indicating significant risk of safety for participants in the study such as: Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third degree AV block)
    * History of familial long QT syndrome or known family history of Torsades de Pointes
    * Cardiac or cardiac repolarization abnormality, including any of the following: History of myocardial infarction (MI), angina pectoris, or coronary artery bypass graft (CABG) within 6 months prior to ICF signature
13. History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study
14. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression
15. Any condition that precludes raised arms position
16. Unmanageable concurrent bladder outflow obstruction or urinary incontinence. Note: participants with bladder outflow obstruction or urinary incontinence, which is manageable and controlled with best available standard of care (incl. pads, drainage) are allowed.
17. Sexually active males unwilling to use a condom during intercourse while taking study treatment and for 14 weeks after stopping study treatment. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner. In addition, male participants must not donate sperm for the time period specified above. If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the ICF

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male prostate cancer patients
Enrollment: 1145 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2027-02-11 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 50 months (estimated final OS analysis)
  rPFS is defined as the time of radiographic progression by Prostate Cancer Working Group 3 (PCWG3)-modified RECIST V1.1 as assessed by blinded independent central review, or death

SECONDARY OUTCOMES:
Overall Survival (OS) (Key Secondary Endpoint) | From date of randomization until date of death from any cause, assessed up to 50 months (estimated final OS analysis)
  OS is defined as time to death for any cause
Prostate-specific antigen 90 (PSA90) response | From date of randomization till 30 days safety fup, assessed up to 50 months (estimated final OS analysis)
  PSA90 response is defined as the proportion of patients who have a more/equal 90% decrease in PSA from baseline, it will be calculated at 12, 24 and 48 months
time to development of mCRPC | From date of randomization till End Of Treatment (EOT) or death, which ever happen first, assessed up to 50 months (estimated final OS analysis)
  Time to development of mCRPC is defined as the time from date of randomization to disease progression despite androgen deprivation therapy (ADT) presenting as either a continuous rise in serum prostate-specific antigen (PSA) levels, the progression of pre existing disease, and/or the appearance of new metastases.
Progression Free Survival (PFS) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to 50 months (estimated final OS analysis)
  PFS is defined as the time from date of randomization to the date of first documented progression by investigator assessment (radiographic progression, clinical progression, PSA progression) or death from any cause, whichever occurs first
second Progression Free Survival (PFS2) | From date of randomization until date of second progression or date of death from any cause, whichever comes first, assessed up to 50 months (estimated final OS analysis)
  PFS2 is defined as time from date of randomization to the first documented progression by investigator assessment (radiographic progression, clinical progression, PSA progression) on next-line therapy or death from any cause, whichever occurs first.
Change in nadir level of PSA lower than 0.2 ng/ml | From date of randomization till 30 days safety fup, whichever occur first, assessed up to 50 months (estimated final OS analysis)
  Proportion of patients with PSA < 0.2 ng/mL at months 12, 24 and 48 months
Time to radiographic soft tissue progression (TTSTP) | From date of randomization until date of soft tissue radiographic progression or date of death from any cause, whichever comes first, assessed up to 50 months (estimated final OS analysis)
  TTSTP is defined as time from randomization to radiographic soft tissue progression per PCWG3-modified RECIST v1.1 (Soft Tissue Rules of Prostate Cancer Working Group modified Response Evaluation Criteria in Solid Tumors Version 1.1) as assessed by Blinded Independent Central Review (BICR)
Time to first symptomatic skeletal event (SSE). | From date of randomization till EOT or death, whichever happens first, assessed up to 50 months (estimated final OS analysis)
  Time to SSE (TTSSE) is defined as date of randomization to the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death from any cause, whichever occurs first
Overall Response Rate (ORR) | From date of randomization till 30 days safety fup, assessed up to 50 months (estimated final OS analysis)
  ORR is defined as the proportion of participants with best overall response of complete response or partial response in soft tissue as per BIRC and according to PCWG3 modified RECIST 1.1
Disease Control Rate (DCR) | From date of randomization till 30 days safety fup, assessed up to 50 months (estimated final OS analysis)
  DCR is defined as the proportion of participants with best overall response of complete response or partial response or Stable disease in soft tissue as per BIRC and according to PCWG3 modified RECIST 1.1
Duration of Response (DOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to 50 months (estimated final OS analysis)
  DOR is defined as the duration of time between the date of first documented response (CR or PR) in soft tissue as per BIRC and according to PCWG3 modified RECIST 1.1, and the date of first documented progression or death due to any cause
Time to Response (TTR) | From date of randomization till 30 days safety fup, assessed up to 50 months (estimated final OS analysis)
  TTR is defined as the time from the date of randomization to the date of first documented response (CR or PR).
Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire | From randomization up till 30 day safety Follow-up or week 48 of long term Follow-up for patients prematurely discontinued, assessed up to 50 months (estimated final OS analysis)
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT-General + the Prostate Cancer Subscale (PCS). The FACT-General (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
European Quality of Life ( EuroQoL) -5 Domain 5 Level Scale (EQ-5D-5L) | From screening up till 30 day safety follow-up or week 48 of long term follow up for patient prematurely discontinued, assessed up to 50 months (estimated final OS analysis)
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.
Brief Pain Inventory-short Form (PBI-SF) | From screening up till 30 day safety follow-up or week 48 of long term follow up for patient prematurely discontinued, assessed up to 50 months (estimated final OS analysis)
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item self report questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.
Number of participants with Treatment Emergent Adverse Events | From randomization till 30 days safety follow-up, assessed up to 50 months (estimated final OS analysis)
  The distribution of adverse events (AE) will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (150):
- United States (69):
  - Mayo Clinic - Arizona Mayo Clinic Hospital, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California San Diego - Moores Cancer Center, La Jolla, California
  - VA Greater LA Healthcare System, Los Angeles, California
  - University of California LA, Los Angeles, California
  - St. Joseph Hospital, Orange, California
  - Univ Cali Irvine ALS Neuromuscular, Orange, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University Medical Center, Palo Alto, California
  - Sansum Clinic, Santa Barbara, California
  - Providence Saint Johns Health Ctr, Santa Monica, California
  - Univ Of Color Anschutz Med Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Georgetown University-Lombardi Cancer Center, Washington D.C., District of Columbia
  - VA Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - University Of Miami, Miami, Florida
  - Miami Cancer Institute at Bapt, Miami, Florida
  - Florida Cancer Affiliates, Panama City, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - The Queens Medical Centre, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Hines VA Hospital, Hines, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University, Indianapolis, Indiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Sidney Kimmel CCC At JH, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Uni Of Michigan Health System, Ann Arbor, Michigan
  - Corewell Health William Beaum Hosp, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Med Ctr, Jackson, Mississippi
  - St. Louis University, St Louis, Missouri
  - VA St Louis Health Care System, St Louis, Missouri
  - Wash U School of Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Urology Cancer Center PC, Omaha, Nebraska
  - University of New Mexico, Albuquerque, New Mexico
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Univ Of Rochester Cancer Ctr, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Univ Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Dallas VA Medical Center, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Univ of Texas Southwest Med Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - UT Health Science Center, Houston, Texas
  - UT Health San Antonio Mays Cancer Center, San Antonio, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onco Hemato Asso of SW Virginia, Roanoke, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Austria (3):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- Canada (6):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (7):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Copenhagen, Denmark
- France (9):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (6):
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Rostock
- Japan (15):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Yamagata
- Netherlands (4):
  - Novartis Investigative Site, Nijmegen, Gelderland
  - Novartis Investigative Site, Maastricht, Limburg
  - Novartis Investigative Site, Delft, South Holland
  - Novartis Investigative Site, Utrecht
- Poland (3):
  - Novartis Investigative Site, Gliwice, Silesian Voivodeship
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (6):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com